CLINICAL TRIAL: NCT06329882
Title: Doxycycline in Combination With Sitagliptin on the Glycemic and Cardiac Indices in Patients With Type 2 Diabetes Mellitus
Brief Title: Doxycycline in Type II Diabetes
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mostafa Bahaa (Other)
Responsible Party: Sponsor-Investigator, Mostafa Bahaa, Teaching assisstant, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14789
Record Dates: First submitted 2024-03-09; First posted 2024-03-26 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Doxycycline

STUDY DESIGN:
Intervention Model Description: open label
Masking Description: open label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): patients were on sitagliptin 100mg /day monotherapy
  Interventions: Drug: Sitagliptin 100mg
- Comparative group (Active Comparator): patients were on sitagliptin 100mg /day monotherapy plus doxycycline 100 mg
  Interventions: Drug: Sitagliptin 100mg; Drug: Doxycyclin

INTERVENTIONS:
Drug: Sitagliptin 100mg — Sitagliptin is used along with diet and exercise and sometimes with other medications to lower blood sugar levels in adults with type 2 diabetes
Drug: Doxycyclin — Doxycycline belongs to the class of medicines known as tetracycline antibiotics. It works by killing bacteria or preventing their growth.
  Arms: Comparative group

SUMMARY:
Type 2 diabetes mellitus (T2DM) is a chronic metabolic disease characterized by hyperglycemia, weight loss, and cardio-metabolic complications. T2DM develops due to the progression of insulin resistance (IR), impairment of insulin insensitivity, and failure of the pancreatic β-cells to release sufficient amount of insulin in response to glucose burden

ELIGIBILITY:
Inclusion Criteria:

* Male or female sex more than 40 years old Newly diagnosed type II diabetes. HbA1c more than 6.5

Exclusion Criteria:

* Patient with chronic kidney disease, hepatic disorders, mental and psychiatric disorders, pregnancy, and lactation

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-30 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Change in glycemic profile | 3 months
  measurement of fasting blood glucose (FBG)
Change in glycemic profile | 3 months
  measurement of glycated hemoglobin

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta Unuversity, Tanta, Egypt